CLINICAL TRIAL: NCT07156734
Title: Does NMES Applied to the Contralateral Uninjured Side Facilitate Voluntary Quadriceps Activation Before and After ACL Surgery?
Brief Title: Effect of Contralateral NMES on Quadriceps Activation After ACL Injury or Surgery
Acronym: ACLQuadAct
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Nicola Maffiuletti, Head Research Group Human Performance Lab, Schulthess Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-00224
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contralateral NMES (Experimental): Participants receive neuromuscular electrical stimulation (NMES) applied to the quadriceps muscle of the contralateral leg while performing voluntary quadriceps contractions on the injured side. Each participant completes two sessions: one after ACL injury and one after ACL reconstruction surgery.
  Interventions: Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Studies in healthy individuals have demonstrated that NMES applied to the quadriceps of one limb induces short-term increases in strength and neural drive in the contralateral homologous muscle. Since these effects have only been observed in healthy individuals, it is essential to investigate whether similar responses occur in ACL patients.

SUMMARY:
A major complication after cruciate ligament injury and surgery is arthrogenic muscle inhibition of the quadriceps, which is characterised by a deficit in voluntary muscle activation in the affected leg. This can hinder rehabilitation processes, lead to impaired knee function, and negatively impact the patients' quality of life. The primary objective of this study is to assess whether voluntary quadriceps activation on the injured side is facilitated by the concomitant application of neuromuscular electrical stimulation (NMES) on the contralateral quadriceps.

DETAILED DESCRIPTION:
The primary objective of this study is to assess whether injured-side voluntary quadriceps activation before and after ACL surgery is facilitated by the concomitant application of NMES on the contralateral quadriceps (uninjured side), in comparison to a control (CTRL) condition that does not involve any contralateral activity (passive rest) and to a voluntary (VOL) condition that involves a maximal voluntary contraction of the contralateral quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACL surgery with semitendinosus tendon autograft in the Schulthess Clinic
* Unilateral and primary ACL injury (with/without diagnoses of additional meniscus injury)

Exclusion Criteria:

* Previous surgery/ligament rupture in injured or uninjured knee or hip
* Severe pain in the uninjured-side quadriceps or knee joint
* Ongoing pregnancy
* BMI >30 kg/m²
* Neuromuscular disease
* Open wounds or tissue injuries on the anterior aspect of the thigh
* Additional rupture of other knee ligaments (posterior cruciate ligament, medial collateral ligament, lateral collateral ligament)
* Implanted metallic/electronic devices (cardiac pacemakers, defibrillators)
* Patients getting a femoralis block (peripheral nerve block) after surgery will be excluded for the post-surgical appointment
* Insufficient language comprehension

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
EMG activity | Data will be collected at two time points: after ACL injury (within two weeks prior to surgery) and following ACL reconstruction (within three days post-surgery).
  EMG data will be recorded from the vastus medialis, vastus lateralis and rectus femoris muscles.

IPD SHARING:
Plan to Share IPD: Undecided